CLINICAL TRIAL: NCT00556504
Title: TCM-700C Phase II Trial The Effects of Adding a Chinese Formulation (TCM-700C) on the Standard Combination Treatment for Patients With Genotype 1 Hepatitis C Infection
Brief Title: The Effects of Adding TCM-700C on the Standard Combination Treatment for Patients With Genotype 1 Hepatitis C Infection
Acronym: TCM-700C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TCM Biotech International Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM-700-01-04
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Hepatitis C
Keywords: add-on treatment; botanical drug; HCV genotype 1; TCM-700C; genotype I
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TCM-700C (Experimental): an add-on drug (2 tablets/t.i.d) to conventional treatment(Peginterferon alfa-2a + ribavirin) of Hepatitis C
  Interventions: Drug: TCM-700C; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Placebo (Placebo Comparator): placebo add on(2 tablets/t.i.d) to conventional treatment(Peginterferon alfa-2a + ribavirin) of Hepatitis C
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin; Drug: Placebo

INTERVENTIONS:
Drug: TCM-700C — An add-on drug to conventional treatment of Hepatitis C
  Arms: TCM-700C
Drug: Peginterferon alfa-2a — conventional treatment of Hepatitis C
  Other Names: Peg-INTRON, Schering-Plough
Drug: Ribavirin — conventional treatment of Hepatitis C
  Other Names: Rebetol, Schering-Plough)
Drug: Placebo — Placebo, without acting ingredient.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of TCM-700C as an add-on treatment to the combination drug therapy (Peginterferon α-2b plus Ribavirin) for patients with genotype 1 chronic hepatitis C infections. This will be demonstrated by a higher sustained virologic response rate, defined as the absence of detectable HCV RNA 24 weeks after the termination of combinational drug treatment, compared with the placebo add-on.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo controlled, parallel-group, Phase 2 study to evaluate the effects of adding a Chinese formulation (TCM-700C) on the standard combination treatment for patients with Genotype 1 hepatitis C infection. Patients were screened within 4 weeks before receive the first study drug dose. Eligible patients at baseline were stratified according to baseline HCV RNA (≤800,000 IU/ml vs >800,000 IU/ml) and randomized with an equal chance to receive either TCM-700C or placebo as an add-on to the combination drug therapy. The combination drug therapy was peginterferon α-2b (PEG-INTRON®, Schering-Plough) 1.5 micrograms/kg once weekly injection for 48 weeks plus oral ribavirin (REBETOL®, Shering-Plough) 1000mg-1200mg daily for 48 weeks. The add-on treatment of TCM-700C or placebo was given 2 tablets thrice daily for 48 weeks.

During the 48 week treatment period and 24 week untreated follow-up, patients were assessed at regular intervals for safety and efficacy at weeks 2, 4, 8, 12, 16 and then every 8 weeks thereafter until study completion. Patients who prematurely discontinued test drug therapy had laboratory examination re-taken on the week patient was discontinued from study.

ELIGIBILITY:
Inclusion Criteria:

* HCV strain confirmed as genotype I;
* Elevated ALT (≥1.5 x upper limit of normal)during last 6 months
* Females of childbearing potential with a negative serum pregnancy test
* Subject must be willing to sign a written informed consent
* Subject must be willing and able to adhere to dose and visit schedule.

Exclusion Criteria:

* Serum AFP levels > 400 ng/ml
* Liver biopsy within 12 months prior to study entry showed liver cirrhosis with METAVIR system fibrosis score of 3-4, or hepatocellular carcinoma (HCC);
* Co-infection with hepatitis B virus (HBV);
* Anti-HIV positive;

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-07; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: I-Sheen Sheen, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: 12 Months location: CGMH clinical ceters
Groups:
- TCM-700C: TCM-700C, an add-on drug to conventional treatment (peginterferon α-2b + ribavirin) of Hepatitis C
  TCM-700C (530mg active ingredient/tablet) : 2 tablets t.i.d for 48 weeks peginterferon α-2b: (1.5 micrograms/kg) once weekly injection for 48 weeks ribavirin: 1000mg-1200mg daily for 48 weeks.
- Placebo: Placebo, an add-on drug to conventional treatment (peginterferon α-2b + ribavirin) of Hepatitis C
  Placebo : 2 tablets t.i.d for 48 weeks peginterferon α-2b: (1.5 micrograms/kg) once weekly injection for 48 weeks ribavirin: 1000mg-1200mg daily for 48 weeks.
Period: Overall Study
Arm/Group | TCM-700C | Placebo
Started | 42 | 42
Intend-to Treat Population | 42 | 42
Safety Population | 41 | 42
Completed | 34 | 33
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- TCM-700C: TCM-700C, an add-on drug to conventional treatment of Hepatitis C
- Placebo: Placebo with convetional treatment for HCV patients
- Total: Total of all reporting groups
Arm/Group | TCM-700C | Placebo | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 42 | 84
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (9.58) | 48.74 (11.52) | 48.67 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 37
  Male | 20 | 27 | 47
Region of Enrollment [Number; unit: participants]
  Taiwan | 42 | 42 | 84
Fibrosis score [Number; unit: participants] — Liver biopsy within 12 months prior to study entry showed liver cirrhosis with METAVIR system fibrosis score
  0 No fibrosis
  1. Stellate enlargement of portal tract but without septa formation
  2. Enlargement of portal tract with rare septa formation
  participants
    Fibrosis score 0 | 0 | 2 | 2
    Fibrosis score 1 | 11 | 21 | 32
    Fibrosis score 2 | 31 | 19 | 50

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR)
Description: SVR is defined as no detectable HCV RNA in serum of patient at Week 72, which is 24 weeks after the termination of combination drug treatment..
  1. A subject is a sustained responder at a given week, if the subject has negative HCV RNA at that week and all the subsequent weeks through Week 72.
  2. If a patient has a missing value between visits, then the last non-missing HCV RNA is carried forward to fill in the missing value.
  3. If the patient's HCV RNA at last visit, Week 72 is missing or above the limit of detection, then the patient is a non-responder, even if all the previous visits from baseline onwards were undetectable.
  Serum HCV RNA will be tested using a commercially available real-time polymerase-chain-reaction (PCR) assay kit (Roche Cobas TaqMan HCV assay kit)
Time Frame: 24 weeks after the termination of combinational drug treatment (up to 72 weeks)
Measure: Number; unit: Number of participants with SVR
Arm/Group | TCM-700C | Placebo
Number analyzed (Participants) | 42 | 42
Number of participants with SVR | 27 | 29

2. Secondary Outcome: Virologic Response
Description: undetectable HCV RNA at the end of combination drug treatment
  Serum HCV RNA will be tested using a commercially available real-time polymerase-chain-reaction (PCR) assay kit (Roche Cobas TaqMan HCV assay kit).
Time Frame: at the end of combination drug treatment (up to 48 weeks)
Measure: Number; unit: participants
Arm/Group | TCM-700C | Placebo
Number analyzed (Participants) | 42 | 42
participants | 34 | 31

3. Secondary Outcome: ALT Response
Description: An ALT response is defined as normalization of ALT at the end of combination drug treatment.
  (ALT normalization is defined as ALT level decreases into within the normal range)
Time Frame: at the end of combination drug treatment (up to 48 weeks)
Measure: Number; unit: participants
Arm/Group | TCM-700C | Placebo
Number analyzed (Participants) | 42 | 42
participants | 32 | 30

4. Secondary Outcome: Sustained ALT Response
Description: a sustained ALT response is defined as sustained normalization of ALT 24 weeks after cessation of combination drug treatment.
Time Frame: 24 weeks after the termination of combinational drug treatment (up to 72 weeks)
Measure: Number; unit: participants
Arm/Group | TCM-700C | Placebo
Number analyzed (Participants) | 42 | 42
participants | 26 | 27

5. Secondary Outcome: Combined ALT and Virologic Response
Description: Combined ALT and virologic response at the end of combination drug treatment.
Time Frame: at the end of combination drug treatment (up to 48 weeks)
Measure: Number; unit: participants
Arm/Group | TCM-700C | Placebo
Number analyzed (Participants) | 42 | 42
participants | 31 | 29

6. Secondary Outcome: Immune Cell Normalization
Description: Normalization of immune cells, CD4, CD8 and NK cells at the end of combination drug treatment
  (Immune cell normalization is defined as return of CD4, CD8 and NK cells to normal range)
Time Frame: at the end of combination drug treatment (up to 48 weeks)
Measure: Number; unit: participants
Arm/Group | TCM-700C | Placebo
Number analyzed (Participants) | 42 | 42
participants
  CD4 | 31 | 27
  CD8 | 36 | 31
  NK cells | 37 | 31

7. Secondary Outcome: Immune Cell Normalization
Description: Normalization of immune cells, CD4, CD8 and NK cells at 24 weeks after cessation of combination drug treatment.
Time Frame: 24 weeks after the termination of combinational drug treatment (up to 72 weeks)
Measure: Number; unit: participants
Arm/Group | TCM-700C | Placebo
Number analyzed (Participants) | 42 | 42
participants
  CD4 | 30 | 25
  CD8 | 34 | 30
  NK cells | 36 | 31

ADVERSE EVENTS:
Time Frame: 72 weeks
Description: Adverse reactions are monitored in all patients who were enrolled and took the study drugs at least one time in the study.
  one patient was excluded from safety population because did not meet the eligibility criteria and did not take any study medication.
Groups:
- TCM-700C (Safety Population): TCM-700C, an add-on drug to conventional treatment(PegIFN plus RBV)of Hepatitis C
- Placebo (Safety Population): Placebo with convetional treatment(PegIFN plus RBV) for HCV patients
Arm/Group | TCM-700C (Safety Population) | Placebo (Safety Population)
Serious Adverse Events (participants affected / at risk) | 9/41 | 6/42
Other Adverse Events (participants affected / at risk) | 41/41 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCM-700C (Safety Population) (N=41) | Placebo (Safety Population) (N=42)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Urinary infection (Infections and infestations) | 2 (2) | 1 (1)
Fever/pain (General disorders) | 2 (2) | 2 (2)
block stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
sinusitis (General disorders) | 0 (0) | 1 (1)
hearing impairment (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Rhinorhea (Endocrine disorders) | 1 (1) | 1 (1)
neuritic depression (Nervous system disorders) | 1 (1) | 0 (0)
lose weight (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TCM-700C (Safety Population) (N=41) | Placebo (Safety Population) (N=42)
Anemia (Blood and lymphatic system disorders) | 8 | 10
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Palpiations (Cardiac disorders) | 3 | 4
Deafness (Ear and labyrinth disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Goitre (Endocrine disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 4 | 0
Conjunctivities (Eye disorders) | 2 | 1
Dry Eye (Eye disorders) | 0 | 2
Eye pain (Eye disorders) | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal distention (Gastrointestinal disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 5 | 6
Apthous stomatits (Gastrointestinal disorders) | 2 | 4
Diarrhea (Gastrointestinal disorders) | 5 | 6
Dry mouth (Gastrointestinal disorders) | 3 | 6
Hemorrhoids (Gastrointestinal disorders) | 1 | 3
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 5 | 8
Peptic ulcer (Gastrointestinal disorders) | 4 | 1
Reflux esophagitis (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 3
Chills (General disorders) | 5 | 2
Malaise (General disorders) | 5 | 8
Pain (General disorders) | 4 | 4
Gallbladder polyp (Hepatobiliary disorders) | 2 | 0
Hepatic steatosis (Hepatobiliary disorders) | 4 | 1
Influenza (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3
Pneumonia (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 4 | 3
Fatigue (General disorders) | 9 | 6
Injection site erythema (General disorders) | 2 | 2
Edema peripheral (General disorders) | 2 | 2
Pyrexia (General disorders) | 17 | 13
Fall (Injury, poisoning and procedural complications) | 2 | 0
Blood uric acid increased (Investigations) | 0 | 3
Hemoglobin decreased (Investigations) | 10 | 9
Neutrophil count decreased (Investigations) | 2 | 3
Weight decreased (Investigations) | 3 | 4
White blood cell count decreased (Investigations) | 4 | 2
Anorexia (Metabolism and nutrition disorders) | 5 | 6
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4
Hyperuricaemi (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2 | 1
Dizziness (Nervous system disorders) | 11 | 8
Headache (Nervous system disorders) | 11 | 4
Hypoesthesia (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 0 | 2
Aggression (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 10 | 8
Mood altered (Psychiatric disorders) | 2 | 2
Dysuria (Renal and urinary disorders) | 1 | 2
Urinary incontinency (Renal and urinary disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 7
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 16
Rash (Skin and subcutaneous tissue disorders) | 8 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 4 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less